CLINICAL TRIAL: NCT05851690
Title: Bilaterally Parallel Elliptic Flap Versus Karydakis Flap in Pilonidal Sinus Disease: A Randomized Controlled Trial
Brief Title: Comparison of Two Different Flap Methods in the Treatment of Pilonidal Sinus Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Umut Fırat Turan, Asst. Prof., Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-16-975
Record Dates: First submitted 2023-04-30; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Pilonidal Sinus
Keywords: Pilonidal sinus disease; Flap; Karydakis; Bilaterally parallel elliptic
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Parallel Elliptic Flap (Active Comparator): Patients operated with the bilateral parallel elliptic flap technique.
  Interventions: Procedure: Surgical treatment of pilonidal sinus disease
- Karydakis Flap (Active Comparator): Patients operated with the karydakis flap technique.
  Interventions: Procedure: Surgical treatment of pilonidal sinus disease

INTERVENTIONS:
Procedure: Surgical treatment of pilonidal sinus disease — Advancement flap techniques in surgical treatment of pilonidal sinus disease.

SUMMARY:
Sacrococcygeal pilonidal sinus disease (PSD) has been defined as a disease characterized by chronic inflammation and recurrent infections caused by the movement of hair toward the gluteal sulcus. This condition is especially seen in young men and negatively affects the quality of life of patients and prevents them from performing their work and school activities. The treatment options for PSD range from the use of antibiotics alone to reconstructed excision with tissue flaps. Although the optimal surgical treatment option remains controversial, expectations from the ideal surgical treatment include low recurrence and postoperative complication rates, early wound healing, short hospital stay, early return to work, and good cosmetic outcomes. The aim of this study was to compare the efficacy of the different flap techniques in the surgical treatment of PSD and evaluate the long-term outcomes of patients.

ELIGIBILITY:
Inclusion Criteria:

* Underwent surgery due to pilonidal sinus disease

Exclusion Criteria:

* Patients with a history of previous pilonidal sinus surgery,
* An acute pilonidal abscess,
* immunodeficiency,
* using immunosuppressive drugs,
* refuse to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Time taken to return to work/school | The patients' return to work ranged from 11 to 49 days.
  Time to return to work in daily life after surgery
Postoperative pain | 1 day
  The pain scores of the patients were determined on the first postoperative day. The Visual Analog Scale (VAS), scored from 1 to 10, was administered to the patients to evaluate their postoperative pain levels.

SECONDARY OUTCOMES:
Length of hospital stay | The patients' length of hospital stay ranged from 1 to 4 days.
  Time to discharge from hospital after surgery
Recurrence of the disease | 43 months
  Recurrence of the disease

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: One year from the date of publication.

REFERENCES:
- [Result] Bi S, Sun K, Chen S, Gu J. Surgical procedures in the pilonidal sinus disease: a systematic review and network meta-analysis. Sci Rep. 2020 Aug 13;10(1):13720. doi: 10.1038/s41598-020-70641-7. PMID 32792519
- [Result] Duman K, Girgin M, Harlak A. Prevalence of sacrococcygeal pilonidal disease in Turkey. Asian J Surg. 2017 Nov;40(6):434-437. doi: 10.1016/j.asjsur.2016.04.001. Epub 2016 May 14. PMID 27188235
- [Result] Johnson EK, Vogel JD, Cowan ML, Feingold DL, Steele SR; Clinical Practice Guidelines Committee of the American Society of Colon and Rectal Surgeons. The American Society of Colon and Rectal Surgeons' Clinical Practice Guidelines for the Management of Pilonidal Disease. Dis Colon Rectum. 2019 Feb;62(2):146-157. doi: 10.1097/DCR.0000000000001237. No abstract available. PMID 30640830
- [Result] Karydakis GE. New approach to the problem of pilonidal sinus. Lancet. 1973 Dec 22;2(7843):1414-5. doi: 10.1016/s0140-6736(73)92803-1. No abstract available. PMID 4128725
- [Result] Iesalnieks I, Ommer A, Herold A, Doll D. German National Guideline on the management of pilonidal disease: update 2020. Langenbecks Arch Surg. 2021 Dec;406(8):2569-2580. doi: 10.1007/s00423-020-02060-1. Epub 2021 May 5. PMID 33950407
- [Result] Yuksel BC, Berkem H, Ozel H, Hengirmen S. A new surgical method of pilonidal sinus treatment: a bilaterally paralel elliptic fascio-cutaneous advancement flap technique. Bratisl Lek Listy. 2012;113(12):728-31. doi: 10.4149/bll_2012_165. PMID 23173633
- [Result] Keshvari A, Keramati MR, Fazeli MS, Kazemeini A, Nouritaromlou MK. Risk factors for complications and recurrence after the Karydakis flap. J Surg Res. 2016 Jul;204(1):55-60. doi: 10.1016/j.jss.2016.04.035. Epub 2016 Apr 23. PMID 27451868
- [Result] Alvandipour M, Zamani MS, Ghorbani M, Charati JY, Karami MY. Comparison of Limberg Flap and Karydakis Flap Surgery for the Treatment of Patients With Pilonidal Sinus Disease: A Single-Blinded Parallel Randomized Study. Ann Coloproctol. 2019 Dec 31;35(6):313-318. doi: 10.3393/ac.2018.09.27. Epub 2019 May 22. PMID 31113167
- [Result] Erkent M, Sahiner IT, Bala M, Kendirci M, Yildirim MB, Topcu R, Bostanoglu S, Dolapci M. Comparison of Primary Midline Closure, Limberg Flap, and Karydakis Flap Techniques in Pilonidal Sinus Surgery. Med Sci Monit. 2018 Dec 11;24:8959-8963. doi: 10.12659/MSM.913248. PMID 30531689
- [Result] Sewefy AM, Hassanen A, Atyia AM, Saleh SK. Karydakis Flap With Compressing Tie-over Interrupted Sutures Without Drain versus Standard Karydakis for Treatment of Sacrococcygeal Pilonidal Sinus Disease. Dis Colon Rectum. 2017 May;60(5):514-520. doi: 10.1097/DCR.0000000000000784. PMID 28383451
- [Result] Al-Khamis A, McCallum I, King PM, Bruce J. Healing by primary versus secondary intention after surgical treatment for pilonidal sinus. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD006213. doi: 10.1002/14651858.CD006213.pub3. PMID 20091589
- [Result] Segre D, Pozzo M, Perinotti R, Roche B; Italian Society of Colorectal Surgery. The treatment of pilonidal disease: guidelines of the Italian Society of Colorectal Surgery (SICCR). Tech Coloproctol. 2015 Oct;19(10):607-13. doi: 10.1007/s10151-015-1369-3. Epub 2015 Sep 16. PMID 26377583
- [Result] Keshvari A, Keramati MR, Fazeli MS, Kazemeini A, Meysamie A, Nouritaromlou MK. Karydakis flap versus excision-only technique in pilonidal disease. J Surg Res. 2015 Sep;198(1):260-6. doi: 10.1016/j.jss.2015.05.039. Epub 2015 May 28. PMID 26094093
- [Result] Tokac M, Dumlu EG, Aydin MS, Yalcin A, Kilic M. Comparison of modified Limberg flap and Karydakis flap operations in pilonidal sinus surgery: prospective randomized study. Int Surg. 2015 May;100(5):870-7. doi: 10.9738/INTSURG-D-14-00213.1. PMID 26011208
- [Result] Arslan K, Said Kokcam S, Koksal H, Turan E, Atay A, Dogru O. Which flap method should be preferred for the treatment of pilonidal sinus? A prospective randomized study. Tech Coloproctol. 2014 Jan;18(1):29-37. doi: 10.1007/s10151-013-0982-2. Epub 2013 Feb 21. PMID 23430349
- [Result] Bali I, Aziret M, Sozen S, Emir S, Erdem H, Cetinkunar S, Irkorucu O. Effectiveness of Limberg and Karydakis flap in recurrent pilonidal sinus disease. Clinics (Sao Paulo). 2015 May;70(5):350-5. doi: 10.6061/clinics/2015(05)08. Epub 2015 May 1. PMID 26039952
- [Result] Ates M, Dirican A, Sarac M, Aslan A, Colak C. Short and long-term results of the Karydakis flap versus the Limberg flap for treating pilonidal sinus disease: a prospective randomized study. Am J Surg. 2011 Nov;202(5):568-73. doi: 10.1016/j.amjsurg.2010.10.021. Epub 2011 Jul 23. PMID 21788003
- [Result] Caliskan M, Kosmaz K, Subasi IE, Acar A, Evren I, Bas G, Atayoglu AT. Comparison of Common Surgical Procedures in Non-complicated Pilonidal Sinus Disease, a 7-Year Follow-Up Trial. World J Surg. 2020 Apr;44(4):1091-1098. doi: 10.1007/s00268-019-05331-1. PMID 31848678
- [Result] Bessa SS. Comparison of short-term results between the modified Karydakis flap and the modified Limberg flap in the management of pilonidal sinus disease: a randomized controlled study. Dis Colon Rectum. 2013 Apr;56(4):491-8. doi: 10.1097/DCR.0b013e31828006f7. PMID 23478617
- [Result] Hull TL, Wu J. Pilonidal disease. Surg Clin North Am. 2002 Dec;82(6):1169-85. doi: 10.1016/s0039-6109(02)00062-2. PMID 12516846
- [Derived] Turan UF, Coban S, Akin T, Berkem H, Yuksel BC, Er S. Bilaterally parallel elliptic flap versus Karydakis flap in primary pilonidal sinus disease: a randomized controlled trial. Int J Colorectal Dis. 2023 Jun 23;38(1):176. doi: 10.1007/s00384-023-04475-w. PMID 37351640